CLINICAL TRIAL: NCT01208311
Title: Acoustic Liver Biopsy in Normals and in Patients With Cirrhosis Using Endoscopic Ultrasound.
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Larry Miller, Principal Investigator, Northwell Health
Other Study IDs: 4539
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Alcoholism; Cirrhosis; Hepatitis c
Keywords: Alcoholic cirrhosis; hepatitis c cirrhosis; cirrhosis
MeSH Terms: conditions — Alcoholism; Fibrosis; Hepatitis C; Liver Cirrhosis, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Hepatitis C Cirrhosis: Patients with Hepatitis C Cirrhosis

SUMMARY:
The purpose of this study is to determine the amount of fibrosis in the liver of hepatitis C patients with advanced fibrosis, using endoscopic ultrasound.

DETAILED DESCRIPTION:
Background: Transabdominal ultrasound cannot be used to quantitate fibrosis in patients with cirrhosis due to variability in the abdominal wall thickness and composition. This variability can be eliminated by using endoscopic ultrasound.

Aim: To determine the amount of fibrosis in the liver of hepatitis C patients with advanced fibrosis, using endoscopic ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* hepatic cirrhosis and hepatitis C and undergoing endoscopy
* Alcoholic liver and undergoing endoscopy
* Normal liver undergoing endoscopy

Exclusion Criteria:

* pregnancy
* Children

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Collect endoscopic ultrasound images form normal subjects, alcoholic liver patients and patients with hepatitis C Cirrhosis.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2004-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Luminosity on ultrasound | Once at the time of the endoscopic ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Larry S Miller, M.D, Principal Investigator — Northwell Health
Locations (1):
- LIJ Medical Center- NSLIJ Health System, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown JJ, Naylor MJ, Yagan N. Imaging of hepatic cirrhosis. Radiology. 1997 Jan;202(1):1-16. doi: 10.1148/radiology.202.1.8988182. No abstract available.
- [Background] Mergo PJ, Ros PR. Imaging of diffuse liver disease. Radiol Clin North Am. 1998 Mar;36(2):365-75. doi: 10.1016/s0033-8389(05)70028-2. PMID 9520988
- [Background] Taylor HM, Ros PR. Hepatic imaging. An overview. Radiol Clin North Am. 1998 Mar;36(2):237-45. doi: 10.1016/s0033-8389(05)70019-1. PMID 9520979
- [Background] Zwiebel WJ. Sonographic diagnosis of diffuse liver disease. Semin Ultrasound CT MR. 1995 Feb;16(1):8-15. doi: 10.1016/0887-2171(95)90011-x. PMID 7718284
- [Background] Aube C, Oberti F, Korali N, Namour MA, Loisel D, Tanguy JY, Valsesia E, Pilette C, Rousselet MC, Bedossa P, Rifflet H, Maiga MY, Penneau-Fontbonne D, Caron C, Cales P. Ultrasonographic diagnosis of hepatic fibrosis or cirrhosis. J Hepatol. 1999 Mar;30(3):472-8. doi: 10.1016/s0168-8278(99)80107-x. PMID 10190731
- [Background] Harbin WP, Robert NJ, Ferrucci JT Jr. Diagnosis of cirrhosis based on regional changes in hepatic morphology: a radiological and pathological analysis. Radiology. 1980 May;135(2):273-83. doi: 10.1148/radiology.135.2.7367613.
- [Background] Hirata M, Akbar SM, Horiike N, Onji M. Noninvasive diagnosis of the degree of hepatic fibrosis using ultrasonography in patients with chronic liver disease due to hepatitis C virus. Eur J Clin Invest. 2001 Jun;31(6):528-35. doi: 10.1046/j.1365-2362.2001.00840.x. PMID 11422403
- [Background] Hultcrantz R, Gabrielsson N. Patients with persistent elevation of aminotransferases: investigation with ultrasonography, radionuclide imaging and liver biopsy. J Intern Med. 1993 Jan;233(1):7-12. doi: 10.1111/j.1365-2796.1993.tb00640.x. PMID 8429291
- [Background] Zheng RQ, Wang QH, Lu MD, Xie SB, Ren J, Su ZZ, Cai YK, Yao JL. Liver fibrosis in chronic viral hepatitis: an ultrasonographic study. World J Gastroenterol. 2003 Nov;9(11):2484-9. doi: 10.3748/wjg.v9.i11.2484. PMID 14606081
- [Result] Andanappa HK, Dai Q, Korimilli A, Panganamamula K, Friedenberg F, Miller L. Acoustic liver biopsy using endoscopic ultrasound. Dig Dis Sci. 2008 Apr;53(4):1078-83. doi: 10.1007/s10620-008-0211-4. Epub 2008 Feb 13. PMID 18270828